CLINICAL TRIAL: NCT03655444
Title: A Prospective Phase I and II Trial of Abemaciclib + Nivolumab in Patients With Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma That Progressed or Recurred Within Six Months After Platinum-based Chemotherapy
Brief Title: Abemaciclib + Nivolumab in Patients With Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma That Progressed or Recurred Within Six Months After Platinum-based Chemotherapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Provider of drug decided to discontinue study.
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201810019
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — abemaciclib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Phase I: Abemaciclib + Nivolumab (Experimental): * Abemaciclib (150 mg) will be administered orally twice per day (with or without food) on Days 1 through 28 of every 4-week cycle
  * Nivolumab 480 mg will be given intravenously (IV) over 30 minutes on Day 1 of every 4-week cycle.
  Interventions: Drug: Abemaciclib; Drug: Nivolumab
- Phase II: Abemaciclib + Nivolumab (Experimental): * Phase II Lead-in: Patients will be treated with abemaciclib monotherapy at the recommended phase II dose (150 mg) on Day -7 through Day -1 prior to starting Cycle 1 with the combination of abemaciclib and nivolumab. Patients will proceed directly from Day -1 to Cycle 1 Day 1 of combination abemaciclib + nivolumab, there is not a Day 0.
  * Patients will be treated with abemaciclib at the RP2D (150 mg) (Days 1 through 28) + nivolumab (480 mg, Day 1) of each 4-week cycle.
  Interventions: Drug: Abemaciclib; Drug: Nivolumab; Procedure: Tumor biopsy; Procedure: Peripheral blood; Other: EORTC QLQ-30

INTERVENTIONS:
Drug: Abemaciclib — Abemaciclib is an investigational agent for this trial and will be supplied by Lilly Oncology, free of charge to the patient.
  Other Names: Verzenio
Drug: Nivolumab — Nivolumab is commercially available
  Other Names: Opdivo
Procedure: Tumor biopsy — * Phase II patients only
  * If the patient consents, fresh tumor tissue will be collected at baseline and then during Cycle 2 (between days 8-22) of abemaciclib and nivolumab.
  Arms: Phase II: Abemaciclib + Nivolumab
Procedure: Peripheral blood — * Phase II patients only
  * Peripheral blood will be collected at baseline, at the end of the Lead In (cycle 1 day 1 prior to treatment), during cycle 2 (between days 8-22), and during cycle 3 (between days 21-28). If patient does not have progression after cycle 3, patient will also have peripheral blood collected at time of progression.
  Arms: Phase II: Abemaciclib + Nivolumab
Other: EORTC QLQ-30 — * Phase II patients only
  * Screening , Cycle 2 D1, Cycle 4 D1, and End of treatment (EOT)
  Arms: Phase II: Abemaciclib + Nivolumab

SUMMARY:
In phase I of the trial, the investigators aim to explore the safety and feasibility of abemaciclib in combination with nivolumab in patients with recurrent/metatstatic head and neck squamous cell carcinoma (RM-HNSCC). A dose de-escalation study design will be used to determine the recommended phase II dose (RP2D) of abemaciclib given with the standard dose of nivolumab.

In phase II of the trial, the investigators aim to determine if abemaciclib and nivolumab will improve the one year survival from 36% (historical comparison with nivolumab) to 60% (abemaciclib + nivolumab) in patients with RM-HNSCC that had progressed or recurred within six months after platinum-based chemotherapy. Patients will be treated with abemaciclib at the recommended phase 2 dose (RP2D) in combination with standard doses of nivolumab. If this aim is met, genome sequencing, bulk and single cell RNAseq, and selected protein expression and deep cellular phenotyping will be performed on tumor tissue and blood obtained before and during treatment with abemaciclib and nivolumab. These biomarker data will be correlated with survival and tumor response to abemaciclib and nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Incurable RM-HNSCC, defined as disease not amenable to cure by surgery and/or radiation therapy (or patient declines or is ineligible for surgery and/or radiation therapy).
* Disease Evaluation:

  * Phase I: evaluable or measurable disease.
  * Phase II: measurable disease, defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm by clinical exam.
* Prior Treatment:

  * Phase I: any number of lines of prior therapy for RM-HNSCC.
  * Phase I: prior therapy with inhibitors of CDK4/6 or PD-L1/PD-1 is acceptable.
  * Phase II: RM-HNSCC that progressed or recurred within six months of platinum-based therapy (given for curable or incurable disease).
  * Phase II: prior therapy with inhibitors of CDK4/6 or PD-L1/PD-1 is not acceptable.
* 18 years of age or older
* Performance status 0-1 (ECOG)
* Adequate blood and organ function as defined:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 8.0 g/dL
  * Total bilirubin ≤ 1.5 x ULN mg/dL
  * AST(SGOT) ≤ 3 x IULN and ALT(SGPT) ≤ 3 x IULN
  * Creatinine ≤ 2 x ULN OR creatinine clearance ≥ 40 mL/min/1.73 m2
  * INR ≤ 1.5 x ULN and PTT ≤ 1.5 x ULN (Patients are allowed to be on anticoagulation)
* Able to swallow oral medication
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) beginning 14 days prior to first dose of abemaciclib, through the dosing period, and for at least 28 days after.
* Signed IRB approved written informed consent document.

Exclusion Criteria:

* Phase II: prior inhibitors of CDK4/6 or PD-L1/PD-1 for treatment of incurable HNSCC.
* Radiation within 14 days of treatment start (patients who received radiotherapy must have completed and fully recovered from the acute side effects of radiotherapy), chemotherapy, targeted or investigational therapy within 21 days of treatment start.
* History of other malignancy ≤ 1 year prior to consent with the exception of completely resected skin carcinoma or other cancers with a low risk of recurrence.
* Ongoing toxicity attributed to prior anti-cancer therapy that is > grade 1, except alopecia or peripheral neuropathy
* Active central nervous system metastases: defined as currently receiving radiation therapy to metastatic CNS disease. Once radiation therapy is completed, patients with CNS disease are eligible if they meet all other criteria for enrollment.
* History of severe allergic reactions attributed to agents used in the study.
* Serious uncontrolled inter-current illness within the 3 months prior to study entry or psychiatric illness/social situations that would limit compliance with study requirements.
* Serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (i.e., interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
* History of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
* Pregnant and/or breastfeeding. Patient must have a negative serum pregnancy test within 7 days of first dose of treatment.
* Active serious autoimmune disease requiring systemic immunosuppression (biologics, prednisone equivalent dose > 20 mg/day).
* Current use of strong CYP3A inhibitors or inducers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Adkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase II: Abemaciclib + Nivolumab: * Phase II Lead-in: Patients will be treated with abemaciclib monotherapy at the recommended phase II dose on Day -7 through Day -1 prior to starting Cycle 1 with the combination of abemaciclib and nivolumab. Patients will proceed directly from Day -1 to Cycle 1 Day 1 of combination abemaciclib + nivolumab, there is not a Day 0.
  * Patients will be treated with abemaciclib at the RP2D (Days 1 through 28) + nivolumab (480 mg, Day 1) of each 4-week cycle.
Period: Overall Study
Arm/Group | Phase I: Abemaciclib + Nivolumab | Phase II: Abemaciclib + Nivolumab
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Abemaciclib + Nivolumab | Phase II: Abemaciclib + Nivolumab | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Median (Full Range); unit: years] | 62 [46 to 76] | 62 [60 to 63] | 62 [46 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Phase I Only: Determine the Recommended Phase 2 Dose of Abemaciclib Combined With a Fixed Dose of Nivolumab
Description: -The RP2D of abemaciclib is defined as the highest dose level at which fewer than 2 patients of a cohort of three patients experience a dose-limiting toxicity (DLT) during the first cycle.
Time Frame: Completion of enrollment to Phase I portion of study (estimated to be 3 months)
Population: Only phase I participants were evaluable for this outcome measure.
Measure: Number; unit: mg twice per day
Arm/Group | Phase I: Abemaciclib + Nivolumab | Phase II: Abemaciclib + Nivolumab
Number analyzed (Participants) | 3 | 0
mg twice per day | 150 |

2. Primary Outcome: Overall Survival (OS) Rate
Description: * OS is defined as the time from the date of treatment to the date of death, censored at the last follow-up otherwise.
  * The mean survival time and standard error were underestimated because the largest observation was censored and the estimation was restricted to the largest event time.
Time Frame: Until death (estimated average of 13 months)
Measure: Mean (Standard Error); unit: months
Groups:
- Phase I and Phase II: Abemaciclib + Nivolumab: * Abemaciclib (150 mg) will be administered orally twice per day (with or without food) on Days 1 through 28 of every 4-week cycle
  * Nivolumab 480 mg will be given intravenously (IV) over 30 minutes on Day 1 of every 4-week cycle.
Arm/Group | Phase I and Phase II: Abemaciclib + Nivolumab
Number analyzed (Participants) | 6
months | 3.689 (0.7281)

3. Secondary Outcome: Phase II Only: Best Overall Tumor Response
Description: * Complete response: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm, Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial response: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.
Time Frame: Through completion of treatment (estimated to be 5 months)
Population: -Phase II patients are the only patients evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Abemaciclib + Nivolumab | Phase II: Abemaciclib + Nivolumab
Number analyzed (Participants) | 0 | 3
Participants |  | 1

4. Secondary Outcome: Phase II Only: Duration of Tumor Response
Description: -The duration of overall response is measured from the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Time Frame: Through completion of treatment (estimated to be 5 months)
Population: Data was not collected for this outcome measure.
Arm/Group | Phase I: Abemaciclib + Nivolumab | Phase II: Abemaciclib + Nivolumab
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Progression-free Survival (PFS)
Description: -PFS is defined as the time from treatment to the date of progression or death, whichever occurs first. The alive patients without progression is censored at the last follow-up.
Time Frame: Through completion of treatment (estimated to be 5 months)
Measure: Mean (Standard Error); unit: months
Arm/Group | Phase I and Phase II: Abemaciclib + Nivolumab
Number analyzed (Participants) | 6
months | 2.82258 (0.64434)

6. Secondary Outcome: Adverse Events (AEs) Associated With the Combination of Abemaciclib and Nivolumab.
Description: -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.
Time Frame: Through 30 days after completion of treatment (estimated to be 6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I and Phase II: Abemaciclib + Nivolumab
Number analyzed (Participants) | 6
Participants
  Anemia | 5
  Hyperthyroidism | 1
  Hypothyroidism | 1
  Constipation | 2
  Diarrhea | 3
  Dry mouth | 1
  Dysphagia | 3
  Mucositis oral | 1
  Nausea | 4
  Vomiting | 3
  Chills | 1
  Edema face | 1
  Fatigue | 5
  Non-cardiac chest pain | 1
  Lung infection | 2
  Thrush | 2
  Vaginal infection | 1
  Alanine aminotransferase increased | 1
  Alkaline phosphatase increased | 2
  Aspartate aminotransferase increased | 3
  Blood bilirubin increased | 1
  Cholesterol high | 1
  Creatinine increased | 6
  Blood bicarbonate decreased | 1
  Lymphocyte count decreased | 6
  Neutrophil count decreased | 2
  Platelet count decreased | 2
  Weight loss | 4
  White blood cell decreased | 2
  Anorexia | 3
  Dehydration | 1
  Hypercalcemia | 2
  Hyperglycemia | 4
  Hyperkalemia | 2
  Hypoalbuminemia | 3
  Hypocalcemia | 1
  Hypoglycemia | 1
  Hypokalemia | 2
  Hypomagnesemia | 1
  Hyponatremia | 3
  Generalized muscle weakness | 1
  Arthritis | 1
  Chest wall pain | 1
  Dizziness | 2
  Dysarthria | 2
  Headache | 1
  Confusion | 1
  Depression | 1
  Acute kidney injury | 1
  Hematuria | 1
  Aspiration | 2
  Cough | 4
  Nasal congestion | 1
  Respiratory failure | 1
  Sore throat | 1
  Pruritus | 2
  Hypertension | 3
  Thromboembolic event | 1

7. Secondary Outcome: Phase II Lead-In Only: Changes in Peripheral Blood Lymphocyte Subsets
Time Frame: Compare before and after one week of abemaciclib monotherapy
Population: The data was not collected for this outcome measure.
Arm/Group | Phase I: Abemaciclib + Nivolumab | Phase II: Abemaciclib + Nivolumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment until 28 days after completion of treatment (median follow-up was 2.8 months)
Arm/Group | Phase I and Phase II: Abemaciclib + Nivolumab
All-Cause Mortality (participants affected / at risk) | 3/6
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I and Phase II: Abemaciclib + Nivolumab (N=6)
Dysphagia (Gastrointestinal disorders) | 1
Lung infection (Infections and infestations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Non cardiac chest pain (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I and Phase II: Abemaciclib + Nivolumab (N=6)
Anemia (Blood and lymphatic system disorders) | 5
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 1
Edema face (General disorders) | 1
Fatigue (General disorders) | 5
Thrush (Infections and infestations) | 2
Vaginal infection (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Cholesterol high (Investigations) | 1
Creatinine increased (Investigations) | 6
Blood bicarbonate decreased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 6
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Investigations) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Generalized muscle weakness (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 3
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT03655444/Prot_SAP_000.pdf